CLINICAL TRIAL: NCT05774743
Title: Use of a Visual Aid in Improving Caregiver Understanding and Recall in Pediatric Anesthesia Consent Process - a Randomized Controlled Trial
Brief Title: Pediatric Anesthesia Consent - Visual Aids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Niveditha Karuppiah, Anesthesiologist, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pediatric Consent
Record Dates: First submitted 2023-02-24; First posted 2023-03-20 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia; Surgery
Keywords: pediatric anesthesia consent
MeSH Terms: interventions — Consent Forms; Audiovisual Aids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Consent (No Intervention): Participants will receive the standard anesthesia consent procedure without the use of the visual aid that is being used in this study.
- Consent with Visual Aid (Experimental): Participants will receive standard anesthesia consent procedure with the use of the visual aid that is being used in this study.
  Interventions: Other: Consent with Visual Aid

INTERVENTIONS:
Other: Consent with Visual Aid — Participants who receive the study intervention will receive the standard anesthesia consent procedure with the addition of the visual aid. The visual aid is a poster with pictorial representations of the information that is verbally communicated to participants during the standard consent process.
  Arms: Consent with Visual Aid

SUMMARY:
Informed consent in pediatric anesthesia is obtained from the caregiver by the anesthesiologist prior to surgery. Studies demonstrate that caregivers often do not fully understand or recall the information (risks and benefits) discussed with them during the consent process. The use of visual aids (pictographs etc.) in the consent process has been studied and found beneficial in increasing recall of the discussion about surgery (appendectomy) and for sedation in the emergency department. The investigators developed posters/pamphlets as visual aids with information about general anesthesia and risks involved to help the caregivers understand the process and risks better when their child comes in for an elective procedure. This randomized controlled trial comparing the recall and satisfaction of the standard consent process with and without the use of the visual aids will help evaluate whether the consent process and caregiver understanding can be improved by using these aids.

DETAILED DESCRIPTION:
The process of consent is unique and challenging in pediatrics as the patients themselves are not able to give their own consent. Instead the consent is given by their caregiver (parent/guardian). The elements of a good consent include - disclosure, comprehension, and voluntary choice.1 To achieve this the physician obtaining consent must clearly communicate and provide the caregivers with the description of the procedures and risks. For the consent process to be successful, it requires the caregiver to understand the information provided to them. The posters will provide the same information on the conduct of a general anesthetic and risks that the anesthesiologist will discuss with the caregivers prior to surgery. The posters will contain pictures and keywords describing the same information. The post consent questionnaire will assess the recall and satisfaction of the caregivers to the consent process.

Various studies have demonstrated the use of visual aids by way of pamphlets, brochures and posters increased patient understanding of medication adherence and the details of surgical procedures.2-5 However, there is no recent data on the use of these aids in the anesthesia consent process, especially in the pediatric population. The investigators aim to develop a visual aid describing the risks of anesthesia to supplement the pediatric consent process. The investigators hope to improve the consent process for pediatric patients and their caregivers and increase caregiver understanding and recall of the risks of general anesthesia. The investigators will include pediatric patients who are undergoing elective surgery under general anesthesia and their caregivers.

Caregivers of pediatric patients who are undergoing elective surgical procedures that require general anesthesia will be recruited to the study and randomized into one of two groups: 1) Group 1 participants will complete the anesthesia consent process as per standard protocol without the use of visual aids. This anesthesia consent process will verbally discuss and explain the type of anesthesia being used, airway management strategies, pain management, and associated risks. The caregivers will then be asked verbally or through writing to answer survey questions which includes caregiver age, sex, education level, occupation, relationship to the patient, and recall of consent process (type of anesthesia, risks involved, etc.). The survey will be administered in the recovery unit after the surgery before discharge from the recovery unit.

Group 2 participants will complete the anesthesia consent process as per standard protocol with the additional use of visual aids (poster that has been attached in Section 2.22). The visual aid will contain a brief note on general anesthesia for elective pediatric surgery and its safety. It will also contain a pictorial representation of the common events and risks involved in receiving a general anesthetic. This anesthesia consent process will verbally and pictorially discuss and explain the type of anesthesia being used, airway management strategies, pain management, and associated risks. The caregivers will then be asked verbally or through writing to answer survey questions which includes caregiver age, sex, education level, occupation, relationship to the patient, and recall of consent process (type of anesthesia, risks involved, etc.). The survey will be administered while the caregivers are in the waiting room during surgery or in the recovery unit after the surgery before discharge from the recovery unit and is expected to take less than 5 minutes to complete. Completion of this survey will end the participants' involvement in this study.

The caregivers will be consented to participate in the study after the anesthesia consent process (but before administration of the caregiver survey) to avoid the risk of recall bias. They will not be made aware of the different methods of consent being administered at the time of anesthesia consent. If the caregiver does not provide consent to participate in this study then the caregiver questionnaire will not be administered and data will not be collected for the purpose of this study. The addition of the visual aids will only enhance the consent process and have the potential for this group of caregiver participants to gain additional information about the anesthesia consent process compared to the standard consent protocol. Thus, since being randomized to the group that would receive the visual aids would not produce any detriment as compared to the standard consent protocol, the study team believes delaying obtaining informed consent to participate in this study until after the anesthesia consent process has been completed is reasonable for this study design.

All statistical analysis will be completed through R Studio version 3.6.0. Descriptive statistics will be reported for baseline characteristic using proportions for categorical variables and means and standard deviations for continuous variables.

If the recall score follows a normal distribution, a two-tailed Student's t-test will be performed to examine the difference in mean recall score between groups otherwise a non-parametric Mann-Whitney U test will be performed. A multivariable linear regression analysis will be performed to estimate correlation coefficients and 95% confidence intervals between baseline characteristics and recall score as a secondary explorative analysis.

ELIGIBILITY:
Inclusion Criteria:

* caregivers of pediatric patients under the age of 18 years old who are undergoing elective surgical procedures (adenoidectomy, tonsillectomy, tympanoplasty, mastoidectomy, strabismus repair, appendectomy, cholecystectomy, herniotomy, circumcision, etc.) requiring a general anesthetic

Exclusion Criteria:Caregivers (study participants) will be excluded from the study if the patient they are a caregiver for meets any of the following criteria:

* having major surgery
* emergency surgery
* ASA (American Society of Anesthesiology) IV and above
* has had previous surgery
* pediatric patients who sign their own consent

Caregivers (study participants) will be excluded if:

* language of communication other than English
* they refuse to provide informed consent

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Difference in the overall recall score | One year
  The primary outcome will be the difference in the overall recall score of risks associated with the surgery and anesthetic (described during the anesthesia consent process) between groups receiving the standard consent process and the standard consent with enhanced visual aid process. The recall score will be calculated using a weight of one unit for each of the fifteen "Common Risks and Events" correctly recalled following the consent process. A mean and standard deviation will be calculated for each group and compared using a two-tailed t-test.
  The scale to be used is the "Common Risks and Events Recall Scale" where each correctly recalled fact presented during the consent process is given a weight of one unit. A higher score indicates better caregiver recall.

SECONDARY OUTCOMES:
Experience of the consent process using Likert scale analysis | One year
  Various factors will be assessed and evaluated as a whole to determine the participant's experience of the consent process and whether the visual aids improved the consent process for participants. Items that will be evaluated and included in the analysis of this outcome include whether participants thought the visual aid improved their understanding of the proposed anesthetic plan (including the risks and benefits), whether they felt that there was sufficient time for the consent process, and whether they felt the consent process was reassuring or threatening. These factors will be evaluated together to form a conclusion regarding this outcome. Each outcome will be evaluated using the same scale of measure (where each participant's response will be given a score using using a Likert scale) and will thus have the same units of measure to allow for aggregate analysis.
Impact of demographic factors on recall score | One year
  The impact of the gender of caregiver, level of caregiver education, and the relationship of caregiver to the patient on recall score will be evaluated through multivariable regression analysis. The recall score will be measured using the "Common Risks and Events Recall Scale" where each correctly recalled fact presented during the consent process is given a weight of one unit. A higher score indicates better caregiver recall.

CONTACTS AND LOCATIONS:
Overall Officials: Niveditha Karuppiah, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenfeld EH, Lopez ME, Yu YR, Justus CA, Borges MM, Mathai RC, Karediya A, Zhang W, Brandt ML. Use of standardized visual aids improves informed consent for appendectomy in children: A randomized control trial. Am J Surg. 2018 Oct;216(4):730-735. doi: 10.1016/j.amjsurg.2018.07.032. Epub 2018 Jul 24. PMID 30060912
- [Background] Li FX, Nah SA, Low Y. Informed consent for emergency surgery--how much do parents truly remember? J Pediatr Surg. 2014 May;49(5):795-7. doi: 10.1016/j.jpedsurg.2014.02.075. Epub 2014 Feb 22. PMID 24851773
- [Background] Lin YK, Yeh YS, Chen CW, Lee WC, Lin CJ, Kuo LC, Shi L. Parental Educational Intervention to Facilitate Informed Consent for Pediatric Procedural Sedation in the Emergency Department: A Parallel-Group Randomized Controlled Trial. Healthcare (Basel). 2022 Nov 23;10(12):2353. doi: 10.3390/healthcare10122353. PMID 36553877
- [Background] Bellolio MF, E Silva LOJ, Puls HA, Hargraves IG, Cabrera D. The research to practice continuum: Development of an evidence-based visual aid to improve informed consent for procedural sedation. J Clin Transl Sci. 2017 Oct;1(5):316-319. doi: 10.1017/cts.2017.303. Epub 2017 Dec 14. PMID 29862058